CLINICAL TRIAL: NCT05738356
Title: Comparison of Three Orthodontic Bonding Systems in White Spot Lesion Development: A Randomized Clinical Trial
Brief Title: Evaluation of White Spot Lesion Development Using 3 Orthodontic Adhesive Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: JUST20220118
Record Dates: First submitted 2023-02-04; First posted 2023-02-22 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: White Spot Lesion
Keywords: Self-etch primer, one step adhesive

STUDY DESIGN:
Intervention Model Description: Three parallel groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator was capturing the images (that were analyzed to measure the outcomes), while a research assistant was saving the images of the patients with coding system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Three-step adhesive (Active Comparator): The orthodontic appliances were bonded to the patients teeth using conventional 3 step adhesive (3M™ Transbond™ XT, 3M Unitek, United States)
  Interventions: Combination Product: Adhesive bonding systems
- Self-etch primer adhesive (Experimental): The orthodontic appliances were bonded to the patients teeth using self-etch primer (3M™ Transbond™ Plus, 3M Unitek, United States).
  Interventions: Combination Product: Adhesive bonding systems
- One-step adhesive system (Experimental): The orthodontic appliances were bonded to the patients teeth using one-step adhesive system (GC Ortho Connect™, GC Orthodontics, Germany)
  Interventions: Combination Product: Adhesive bonding systems

INTERVENTIONS:
Combination Product: Adhesive bonding systems — Three different adhesive bonding systems were used; one system per group

SUMMARY:
The gaol of this randomized clinical trial was to compare the effect of self-etching primer bonding system and one step adhesive bonding system on the development of white spot lesions (WSLs) during fixed orthodontic therapy in comparison with the conventional 3 step bonding system.

All participants will be bonded with similar fixed orthodontic appliances using each type of adhesives for the assigned group. WSLs will be monitored during the orthodontic treatment

DETAILED DESCRIPTION:
Objectives: The objective of this clinical trial was to compare the effect of self-etching primer bonding system and one step adhesive bonding system on the development of WSLs during fixed orthodontic therapy in comparison with the conventional 3 step bonding system.

Materials and Methods: Seventy five patients were randomly allocated into 3 groups (Group 1, conventional bonding system, n=25; Group 2, self-etch primer n=25; Group 3, primer mixed with the adhesive composite n=25). Quantitative light-induced fluorescence (QLF) was used to quantify WSL parameters. Images were captured and then analyzed before treatment; 2 months and 4 months after bond-up. Lesion area (Pixels), mean fluorescence loss (∆F) and the number of newly developed WSLs were compared within and between the 3 groups. The significance level was set at P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients from both sexes aged 17 - 25 years
* Mild-to-moderate crowding (≤5 mm)
* Optimum oral hygiene
* Maximum of 3 restored teeth
* Absence of defective enamel formation in the form of hypocalcification or hypoplasia
* No salivary gland diseases.

Exclusion Criteria:

* Patients with poor oral hygiene
* Heavily restored teeth
* Sever crowding
* Presence of systemic disease that may affect salivary glands or the ability to brush their teeth properly.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Average lesion fluorescence loss (ΔF%) | 4 months
  It reflects mineral loss from tooth surface (in percent)
surface area of WSL | 4 months
  Area of mineral loss measured in pixels
Incidence of WSL | 4 months
  Number of newly developed WSLs

SECONDARY OUTCOMES:
Maximum lesion fluorescence loss (ΔFMAX%) | 4 months
  It reflects the deepest area of the WSL (in percent)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Al-Khateeb, PhD, Principal Investigator — Faculty of Dentistry/Jordan University of Science and Technology
Locations (1):
- Postgraduate Dental Teaching Clinics/JUST, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request

REFERENCES:
- [Background] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Background] Mohammed RE, Abass S, Abubakr NH, Mohammed ZM. Comparing orthodontic bond failures of light-cured composite resin with chemical-cured composite resin: A 12-month clinical trial. Am J Orthod Dentofacial Orthop. 2016 Aug;150(2):290-4. doi: 10.1016/j.ajodo.2016.02.013. PMID 27476362
- [Background] BUONOCORE MG. A simple method of increasing the adhesion of acrylic filling materials to enamel surfaces. J Dent Res. 1955 Dec;34(6):849-53. doi: 10.1177/00220345550340060801. No abstract available. PMID 13271655
- [Background] Frazier MC, Southard TE, Doster PM. Prevention of enamel demineralization during orthodontic treatment: an in vitro study using pit and fissure sealants. Am J Orthod Dentofacial Orthop. 1996 Nov;110(5):459-65. doi: 10.1016/s0889-5406(96)70050-1. PMID 8922502
- [Background] Miller CC, Burnside G, Higham SM, Flannigan NL. Quantitative Light-induced Fluorescence-Digital as an oral hygiene evaluation tool to assess plaque accumulation and enamel demineralization in orthodontics. Angle Orthod. 2016 Nov;86(6):991-997. doi: 10.2319/092415-648.1. Epub 2016 Mar 23. PMID 27007753
- [Background] Bishara SE, Ajlouni R, Laffoon JF, Warren JJ. Comparison of shear bond strength of two self-etch primer/adhesive systems. Angle Orthod. 2006 Jan;76(1):123-6. doi: 10.1043/0003-3219(2006)076[0123:COSBSO]2.0.CO;2. PMID 16448281
- [Background] Elkalza, A., Mostafa, D. (2018). 'Laboratory evaluation of shear bond strength of three different bonding systems for orthodontic brackets', Egyptian Orthodontic Journal, 53(June 2018), pp. 55-60. doi: 10.21608/eos.2018.77121
- [Background] Choi A, Yoo KH, Yoon SY, Park BS, Kim IR, Kim YI. Anti-Microbial and Remineralizing Properties of Self-Adhesive Orthodontic Resin Containing Mesoporous Bioactive Glass. Materials (Basel). 2021 Jun 25;14(13):3550. doi: 10.3390/ma14133550. PMID 34202013
- [Background] Bishara SE, Gordan VV, VonWald L, Olson ME. Effect of an acidic primer on shear bond strength of orthodontic brackets. Am J Orthod Dentofacial Orthop. 1998 Sep;114(3):243-7. doi: 10.1016/s0889-5406(98)70205-7. PMID 9743128
- [Background] Bishara SE, VonWald L, Laffoon JF, Warren JJ. Effect of a self-etch primer/adhesive on the shear bond strength of orthodontic brackets. Am J Orthod Dentofacial Orthop. 2001 Jun;119(6):621-4. doi: 10.1067/mod.2001.113269. PMID 11395706
- [Background] Montasser MA, El-Wassefy NA, Taha M. In vitro study of the potential protection of sound enamel against demineralization. Prog Orthod. 2015;16:12. doi: 10.1186/s40510-015-0080-2. Epub 2015 May 22. PMID 26061985
- [Background] Paschos E, Rosenbeck KA, Huth KC, Rudzki I, Wichelhaus A, Kunzelmann KH. Evaluation of the effect of bracket-periphery treatment on prevention of enamel demineralization by consecutive muCT scans. Clin Oral Investig. 2015 Jul;19(6):1519-26. doi: 10.1007/s00784-014-1351-x. Epub 2014 Nov 14. PMID 25391496
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Albhaisi Z, Al-Khateeb SN, Abu Alhaija ES. Enamel demineralization during clear aligner orthodontic treatment compared with fixed appliance therapy, evaluated with quantitative light-induced fluorescence: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2020 May;157(5):594-601. doi: 10.1016/j.ajodo.2020.01.004. PMID 32354432
- [Background] Al-Khateeb SN, Tarazi SJ, Al Maaitah EF, Al-Batayneh OB, Abu Alhaija ES. Does acid etching enhance remineralisation of arrested white spot lesions? Eur Arch Paediatr Dent. 2014 Dec;15(6):413-9. doi: 10.1007/s40368-014-0131-2. Epub 2014 Jun 21. PMID 24952017
- [Background] Houston WJ. The analysis of errors in orthodontic measurements. Am J Orthod. 1983 May;83(5):382-90. doi: 10.1016/0002-9416(83)90322-6. PMID 6573846
- [Background] Artun J, Brobakken BO. Prevalence of carious white spots after orthodontic treatment with multibonded appliances. Eur J Orthod. 1986 Nov;8(4):229-34. doi: 10.1093/ejo/8.4.229. No abstract available. PMID 3466795
- [Background] Julien KC, Buschang PH, Campbell PM. Prevalence of white spot lesion formation during orthodontic treatment. Angle Orthod. 2013 Jul;83(4):641-7. doi: 10.2319/071712-584.1. Epub 2013 Jan 4. PMID 23289733
- [Background] Brown MD, Campbell PM, Schneiderman ED, Buschang PH. A practice-based evaluation of the prevalence and predisposing etiology of white spot lesions. Angle Orthod. 2016 Mar;86(2):181-6. doi: 10.2319/041515-249.1. Epub 2015 Aug 4. PMID 26241805
- [Background] Paschos E, Kleinschrodt T, Clementino-Luedemann T, Huth KC, Hickel R, Kunzelmann KH, Rudzki-Janson I. Effect of different bonding agents on prevention of enamel demineralization around orthodontic brackets. Am J Orthod Dentofacial Orthop. 2009 May;135(5):603-12. doi: 10.1016/j.ajodo.2007.11.028. PMID 19409343
- [Background] Visel D, Jacker T, Jost-Brinkmann PG, Prager TM. Demineralization adjacent to orthodontic brackets after application of conventional and self-etching primer systems. J Orofac Orthop. 2014 Sep;75(5):358-73. doi: 10.1007/s00056-014-0233-9. Epub 2014 Aug 28. PMID 25158949
- [Background] Rasmussen MJ, Togrye C, Trojan TM, Tantbirojn D, Versluis A. Post-gel shrinkage, elastic modulus, and stress generated by orthodontic adhesives. Angle Orthod. 2020 Mar;90(2):278-284. doi: 10.2319/032719-233.1. Epub 2019 Sep 23. PMID 31545075
- [Background] Ogaard B, Rolla G, Arends J. Orthodontic appliances and enamel demineralization. Part 1. Lesion development. Am J Orthod Dentofacial Orthop. 1988 Jul;94(1):68-73. doi: 10.1016/0889-5406(88)90453-2. PMID 3164585
- [Background] Boersma JG, van der Veen MH, Lagerweij MD, Bokhout B, Prahl-Andersen B. Caries prevalence measured with QLF after treatment with fixed orthodontic appliances: influencing factors. Caries Res. 2005 Jan-Feb;39(1):41-7. doi: 10.1159/000081655. PMID 15591733
- [Background] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Background] Ghiz MA, Ngan P, Kao E, Martin C, Gunel E. Effects of sealant and self-etching primer on enamel decalcification. Part II: an in-vivo study. Am J Orthod Dentofacial Orthop. 2009 Feb;135(2):206-13. doi: 10.1016/j.ajodo.2007.02.060. PMID 19201328
- [Background] Ogaard B. Prevalence of white spot lesions in 19-year-olds: a study on untreated and orthodontically treated persons 5 years after treatment. Am J Orthod Dentofacial Orthop. 1989 Nov;96(5):423-7. doi: 10.1016/0889-5406(89)90327-2. PMID 2816842
- [Background] Donly KJ, Ruiz M. In vitro demineralization inhibition of enamel caries utilizing an unfilled resin. Clin Prev Dent. 1992 Nov-Dec;14(6):22-4. PMID 1298574
- [Background] Cal-Neto JP, Miguel JA. Scanning electron microscopy evaluation of the bonding mechanism of a self-etching primer on enamel. Angle Orthod. 2006 Jan;76(1):132-6. doi: 10.1043/0003-3219(2006)076[0132:SEMEOT]2.0.CO;2. PMID 16448283
- See also: Randomization App — http://www.random.org/sequences/.